CLINICAL TRIAL: NCT01253239
Title: A Retrospective Evaluation Comparing Post Operative Visual Outcomes in Patients Implanted With the TECNIS IOL in Both Eyes Versus the ReZoom IOL in One Eye and TECNIS IOL in the Opposite Eye
Brief Title: Evaluation the TECNIS IOL in Both Eyes VS the ReZoom IOL in One and TECNIS IOL in the Opposite
Status: Completed | Type: Observational
Sponsor: Frank A. Bucci, Jr., M.D. (Other)
Responsible Party: Sponsor-Investigator, Frank A. Bucci, Jr., M.D., Principal Investigator, Bucci Laser Vision Institute
Organization: Bucci Laser Vision Institute (Other)
Other Study IDs: TECNIS-ReZoom-2010
Record Dates: First submitted 2010-11-29; First posted 2010-12-03 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Cataract
Keywords: Visual outcomes; Patient satisfaction
MeSH Terms: conditions — Cataract; Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- TECNIS/ReZoom: Patients who received a TECNIS multifocal IOL in one eye and a ReZoom multifocal IOL in the opposite eye.
- TECNIS/TECNIS: Patients who received TECNIS multifocal IOLs in both eyes

SUMMARY:
The purpose of this study is to evaluate the visual performance of two cohorts of patients who received multifocal intraocular lenses following cataract and clear lens extraction surgeries. Comparing visual outcomes of patients who were implanted with TECNIS Multifocal IOLs in both eyes versus patients implanted with TECNIS Multifocal in one eye and ReZoom Multifocal IOL in the opposite eye.

DETAILED DESCRIPTION:
Stable post operative cataract and clear lens extraction patients who have been implanted with either the TECNIS Multifocal IOL in both eyes or TECNIS Multifocal IOL in one eye and theReZoom Multifocal IOL in the opposite eye.

Study Design-A retrospective chart review to collect visual outcomes to determine lens performance. Patient satisfaction questionnaire will be administered to determine spectacle independence.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone surgery and received either the TECNIS Multifocal Intraocular lens in one eye and the ReZoom Multifocal Intraocular lens in the other will be evaluated. Males and Females with ages ranging from 42 years to 86 years old.

Exclusion Criteria:

* Patients who have subsequently developed any visual limiting problems (e.g. corneal, retinal, infection) which could potentially limit their post operative visual potential.

Ages: 42 Years to 86 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Stable post operative cataract and clear lens extraction patients who have been implanted with either the TECNIS multifocal IOLs in both eyes or TECNIS multifocal IOL in one eye and the ReZoom in the opposite eye
Sampling Method: Non-Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2010-11; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Uncorrected visual acuity at distance and near | Six months

SECONDARY OUTCOMES:
Patients Satisfaction | Six months

CONTACTS AND LOCATIONS:
Overall Officials: Frank A Bucci, Jr., MD, Principal Investigator — Bucci Laser Vision Institute
Locations (1):
- Bucci Laser Vision Institute, Wilkes-Barre, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided